CLINICAL TRIAL: NCT02369484
Title: Afatinib in Pretreated Patients With Advanced NSCLC Harbouring HER2 Exon 20 Mutations
Brief Title: Afatinib in NSCLC With HER2 Mutation
Acronym: NICHE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 7-14; 2014-005098-35 (EudraCT Number); 1200.230 (Other: Boehringer Ingelheim); SNCTP000001674 (Registry Identifier: Swiss National Clinical Trials Portal (SNCTP))
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: NSCLC
Keywords: Stage IIIb/ IV NSCLC harbouring HER2 exon 20 mutations
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Afatinib (Other): Afatinib 40 mg p.o./day until tumour progression or lack of tolerability
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — 40mg p.o./ day until documented progression or unacceptable toxicity
  Other Names: Giotrif; BIBW 2992

SUMMARY:
The purpose of this study is to investigate the control of disease in pretreated patients with advanced non small cell lung cancer (NSCLC) harbouring HER2 exon 20 mutations as well as the safety and tolerability (how severe the side effects are) of the treatment with afatinib.

DETAILED DESCRIPTION:
Previous clinical studies of NSCLC have shown that patients with tumors harboring specific gene mutations (changes) in the epithelial growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) showed better results after treatment with tyrosine kinase inhibitors (TKI), like afatinib (tradename Giotrif®) , compared with classical treatment with chemotherapy. The treatment with TKI has become a new standard-of-care for patient with advanced lung cancer and EGFR or ALK changes. Several novel mutations, which are candidates as targets for specific medication have been discovered. Human epidermal growth factor 2 (HER2, erbB-2/neu) is a protein of the so called ErbB family (including HER2 [ErbB2], ErbB3 and ErbB4). These proteins are involved in the growth and spread of cancer cells. Mutations in HER2 are found in about 2% of the NSCLC.

Afatinib works by blocking the activity of the ErbB family proteins and can inhibit growth and spread of cancer cells. Afatinib is approved by the European and the Swiss Medicines Agencies for the treatment of adult patients with a specific type of cancer of the lung (non-small cell lung cancer) that is identified by a change (mutation) in the gene for EGFR as first treatment or if prior chemotherapy treatment has been insufficient.

A total of 22 patients from centers around Europe are expected to be enrolled in this study over a period of 24 months.

All patients will be treated in the same way. The study will take approximately 40 months to be completed.

This clinical trial is conducted according to the applicable national laws and international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non small cell lung cancer
* Stage IIIB (non amenable to curative-intent multimodal treatment) or IV NSCLC, according to 7th TNM classification.
* Contrast-enhanced CT of thorax and upper abdomen (incl. liver, kidney, adrenals);
* brain MRI or CT within 28 days before the date of enrolment.
* Non-predominant squamous subtype (<50% squamous cells).
* Previous treatment with a platinum based chemotherapy for advanced disease; or Disease relapse or progression within <6 months after adjuvant platinum based chemotherapy, or (definitive) platinum-based chemo(radio)therapy for stage I-III NSCLC
* Measurable or evaluable disease (according to RECIST 1.1 criteria). Not eligible: patients with only one measurable or evaluable tumour lesion which was resected or irradiated prior to enrolment.
* Locally documented HER2 mutation
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Life expectancy >3 months.
* Adequate haematological function:
* WBC ≥ 2000/μL
* haemoglobin ≥ 9 g/dL
* neutrophils count ≥1.5×109/L
* platelet count ≥ 100 × 109/L
* Adequate liver function:
* Total bilirubin ≤ 1.5 × ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* ALT < 2.5 × ULN
* AST < 2.5 × ULN
* GGT < 2.5 × ULN.
* Adequate renal function: Calculated creatinine clearance ≥ 45mL/min (Cockroft-Gault)
* Patient capable of proper therapeutic compliance, and accessible for correct followup.
* Women of childbearing potential (< 1 year without menstruation or < 2 years without menstruation following chemotherapy) must have a negative serum or urine pregnancy test within 7 days before beginning trial treatment.
* Sexually active men and women of childbearing potential must use an effective contraceptive method (two barrier methods or a barrier method plus a hormonal method) during the trial treatment and for a period of at least 28 days following the last administration of trial drug.
* Recovered from any previous therapy related toxicity to ≤Grade 1 at date of enrolment (except for recovery to ≤Grade 2 of alopecia, fatigue, creatinine increased, lack of appetite as well as stable sensory neuropathy)
* Written Informed Consent (IC) for trial treatment must be signed and dated by the patient and the investigator prior to any trial-related intervention.
* Tumour block available for central review of HER2 mutation status.

Exclusion Criteria:

* Patient with mixed small-cell and non-small-cell histologic features
* Uncontrolled lepto-meningeal metastatic disease. Radiotherapy-treated or asymptomatic brain metastases are allowed (no systematic screening). Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids or have been on stable dose of corticosteroids for at least 4 weeks before starting trial treatment. Any symptoms attributed to brain metastases must be stable for at least 4 weeks before date of enrolment.
* Previous treatment with HER2 targeted antibody or tyrosine kinase inhibitor including afatinib.
* Major surgery within 4 weeks before starting trial treatment or scheduled for surgery during the projected course of the trial.
* Patient who has had in the past 3 years any previous or concomitant malignancy EXCEPT adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, in situ ductal carcinoma of the breast.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of III or IV (see Table 2 below), unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to enrolment.
* Patient with other serious diseases or clinical conditions, including but not limited to uncontrolled active infection and any other serious underlying medical processes that could affect the patient's capacity to participate in the trial.
* Known HIV, active Hepatitis B or Hepatitis C infection (screening not required).
* Known or suspected hypersensitivity to afatinib or any of its excipients.
* Interstitial lung disease or pulmonary fibrosis.
* Women who are pregnant or in the period of lactation.
* Patients with any concurrent systemic anticancer therapy.
* Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the trial drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhea, malabsorption.
* Patient who received treatment with an investigational drug agent during the 3 weeks before enrolment in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solange Peters, MD-PhD, Study Chair — Centre Hospitalier Universitaire Vaudois (CHUV); Lausanne, Switzerland; Rafal Dziadziuszko, MD, Study Chair — Medical University of Gdansk, Gdansk, Poland
Locations (5):
- Universitätsklinikum Köln, Cologne, Germany
- NKI-AVL, Amsterdam, Netherlands
- Vall d'Hebron University Hospital, Barcelona, Spain
- Switzerland (2):
  - CHUV, Lausanne
  - USZ, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazieres J, Peters S, Lepage B, Cortot AB, Barlesi F, Beau-Faller M, Besse B, Blons H, Mansuet-Lupo A, Urban T, Moro-Sibilot D, Dansin E, Chouaid C, Wislez M, Diebold J, Felip E, Rouquette I, Milia JD, Gautschi O. Lung cancer that harbors an HER2 mutation: epidemiologic characteristics and therapeutic perspectives. J Clin Oncol. 2013 Jun 1;31(16):1997-2003. doi: 10.1200/JCO.2012.45.6095. Epub 2013 Apr 22. PMID 23610105
- [Background] De Greve J, Teugels E, Geers C, Decoster L, Galdermans D, De Mey J, Everaert H, Umelo I, In't Veld P, Schallier D. Clinical activity of afatinib (BIBW 2992) in patients with lung adenocarcinoma with mutations in the kinase domain of HER2/neu. Lung Cancer. 2012 Apr;76(1):123-7. doi: 10.1016/j.lungcan.2012.01.008. Epub 2012 Feb 10. PMID 22325357
- [Background] Tomizawa K, Suda K, Onozato R, Kosaka T, Endoh H, Sekido Y, Shigematsu H, Kuwano H, Yatabe Y, Mitsudomi T. Prognostic and predictive implications of HER2/ERBB2/neu gene mutations in lung cancers. Lung Cancer. 2011 Oct;74(1):139-44. doi: 10.1016/j.lungcan.2011.01.014. Epub 2011 Feb 25. PMID 21353324
- See also: Sponsor — http://www.etop-eu.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ETOP/7-14 NICHE trial was activated in December 2014. The first patient was enrolled on September 2015 while the last one on August 2016, before accrual was suspended in October 2016. Patients were enrolled in 3 centers (Netherlands Cancer Institute of Amsterdam, Vall d' Herbon Univesity Hospital (Spain) and Universitatsklinikum Koln (Germany)).
Pre-assignment Details: All 13 patients eligible for enrollment received treatment
Period: Overall Study
Arm/Group | Afatinib
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Afatinib
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] — Age of patient at enrollment
  years | 59 [39 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 7
  Germany | 3
  Spain | 3
Smoking history [Count of Participants; unit: Participants]
  Current | 1
  Former | 4
  Never | 8
ECOG Performance status [Count of Participants; unit: Participants] — PS 0: Fully active, able to carry on all pre-disease performance without restriction.
  PS 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  PS 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  PS 3: Capable of only limited self care, confined to bed or chair more than 50% of waking hours.
  PS 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  Participants
    0 | 7
    1 | 4
    2 | 2
T parameter [Count of Participants; unit: Participants] — Primary tumor (T)
  TX: Main tumor cannot be measured. T0: Main tumor cannot be found. T1, T2, T3, T4: Refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T1b | 1
    T2a | 3
    T3 | 3
    T4 | 6
N parameter [Count of Participants; unit: Participants] — Regional lymph nodes (N)
  NX: Cancer in nearby lymph nodes cannot be measured. N0: There is no cancer in nearby lymph nodes. N1, N2, N3: Refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer.
  Participants
    N0 | 5
    N2 | 3
    N3 | 5
M parameter [Count of Participants; unit: Participants] — Distant metastasis (M)
  MX: Metastasis cannot be measured. M0: Cancer has not spread to other parts of the body. M1: Cancer has spread to other parts of the body.
  Participants
    M0 | 1
    M1a | 6
    M1b | 6
TNM staging [Count of Participants; unit: Participants] — The TNM system is the most widely used cancer staging system.
  In the TNM system:
  The T refers to the size and extent of the main tumor. The main tumor is usually called the primary tumor.
  The N refers to the the number of nearby lymph nodes that have cancer. The M refers to whether the cancer has metastasized. This means that the cancer has spread from the primary tumor to other parts of the body.
  When your cancer is described by the TNM system, there will be numbers after each letter that give more details about the cancer-for example, T1N0MX or T3N1M0.
  Participants
    T1b-N3-M1b | 1
    T2a-N0-M1a | 1
    T2a-N2-M1b | 1
    T2a-N3-M1b | 1
    T3-N0-M1b | 1
    T3-N2-M1a | 1
    T3-N3-M1b | 1
    T4-N0-M1a | 3
    T4-N2-M0 | 1
    T4-N3-M1a | 1
    T4-N3-M1b | 1
Type of prior platinum treatment [Count of Participants; unit: Participants]
  Adjuvant | 2
  Advanced disease | 11

OUTCOME MEASURES:

1. Primary Outcome: Disease Control (Defined as Complete or Partial Response, or Disease Stabilisation Lasting at Least 12 Weeks)
Description: Disease control (DC) is defined as complete or partial response, or disease stabilisation lasting at least 12 weeks.
  Disease control will be determined using RECIST 1.1 criteria:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
  Progression (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum recorded on the trial. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions denotes disease progression.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters recorded on the trial.
Time Frame: at interim (after the first 9 pts have been followed for 12 weeks) & final analysis (approx. 40 months after inclusion of first pt)
Population: The statistical design of the trial, included an interim efficacy analysis to be performed as soon as the 12-week status of the first 9 patients was available. So, the interim analysis was performed but up to then 13 patients have been enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib
Number analyzed (Participants) | 13
Participants
  Analysis of all enrolled patients (N=13): DC at 12 weeks- "Yes" | 7
  Analysis of all enrolled patients (N=13): DC at 12 weeks- "No" | 6
  Interim analysis patients (N=9): number analyzed (Participants) | 9
  Interim analysis patients (N=9): DC at 12 weeks- "Yes" | 4
  Interim analysis patients (N=9): DC at 12 weeks- "No" | 5

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from date of enrollment until documented progression or death, if progression is not documented. Censoring will occur at the last tumor assessment only if patients is lost to follow-up
Time Frame: Time assessed from the date of enrolment until documented progression or death (max 36 months)
Population: All patients enrolled up to trial termination
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Afatinib
Number analyzed (Participants) | 13
weeks | 15.9 [6.0 to 35.4]

3. Secondary Outcome: Objective Response
Description: Objective response is defined as best overall response (CR or PR) across all assessment time-points during the period from enrollment to termination of trial treatment. Objective response to afatinib treatment will be determined using RECIST 1.1 criteria:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
  Progression (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum recorded on the trial. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions denotes disease progression.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters recorded on the trial.
Time Frame: Assessed across all time-points during the period from enrolment to termination of trial treatment (max. 36 months)
Population: All patients enrolled in the trial up to trial termination. From the total of 13 patients, one patient had only one tumor assessment and was classified as "Non-Evaluable", since she cannot be accounted for the Objective Response rate.
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib
Number analyzed (Participants) | 13
Participants
  Objective response (CR or PR) | 1
  Stable disease | 6
  Progression disease | 5
  Non-evaluable | 1

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from the date of enrollment until death from any cause. Censoring will occur at the last follow-up.
Time Frame: Time assessed from the date of enrolment until death (max 36 months)
Population: All patients enrolled in the trial up to trial termination
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Afatinib
Number analyzed (Participants) | 13
weeks | 56.0 [16.3 to 100]

5. Secondary Outcome: Toxicities of Treatment
Description: Adverse events classified according to NCI CTCAE version 4.
Time Frame: Assessed from the date of informed consent until 90 days after the final dose of afatinib (max 18 months).
Population: All patients enrolled in the trial up to trial termination
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib
Number analyzed (Participants) | 13
Participants
  Experienced AE/SAE | 13
  No AE/SAE | 0

ADVERSE EVENTS:
Time Frame: From the date of informed consent until 90 days after the final dose of afatinib (max 18 months).
Arm/Group | Afatinib
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=13)
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=13)
Diarrhea (Gastrointestinal disorders) | 11
Mucositis oral (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3
Paronyclia (Infections and infestations) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Other (Skin and subcutaneous tissue disorders) | 2
Bladder infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary track infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Other (tonsillitis) (Infections and infestations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Flu like symptoms (General disorders) | 2
Non-cardiac chest (General disorders) | 2
Malaise (General disorders) | 1
GGT increased (Investigations) | 2
Asparate aminotransferase increased (Investigations) | 1
Creatine increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight loss (Investigations) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Arthalgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Other (paraplegia from Th4)) (Nervous system disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary track obstruction (Renal and urinary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Ventricular arrhythmia (Cardiac disorders) | 1
Dry eye (Eye disorders) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2014-12-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT02369484/Prot_001.pdf
  • Statistical Analysis Plan (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT02369484/SAP_000.pdf
  • Informed Consent Form (2014-12-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT02369484/ICF_002.pdf